CLINICAL TRIAL: NCT06201936
Title: Evaluation of Preexisting Information Regarding Neuroaxial Procedures for Labour Analgesia
Brief Title: EPIDURAL- Evaluation of Preexisting Information Regarding Neuroaxial Procedures for Labour Analgesia
Acronym: EPIDURAL
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Consultant, Goethe University
Other Study IDs: 2023-1XXX
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Neuroaxial Analgesia Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Preliminary information on neuroaxial procedures — Pre-existing information of pregnant women on neuroaxial pain-relieving procedures for childbirth and their informative sources

SUMMARY:
The aim of this research project is to anonymously survey pregnant patients before the anaesthesiological consultation about their prior knowledge of planned neuroaxial procedures in the context of childbirth by conducting an online survey and to evaluate the sources of that information.

DETAILED DESCRIPTION:
Within labour and delivery, neuroaxial anaesthesia (peridural or spinal anaesthesia) is commonly used in accordance with clinical practice guidelines. However, from a professional perspective, there are still questionable and incorrect statements about possible complications and side effects that cannot be justified medically. In an increasingly technological and networked society, the dissemination of medical information via various sources of information poses a potentially serious problem in terms of disinformation, and the correct classification of information is becoming more and more difficult.

Anaesthesiologists are increasingly confronted with consultations in which, in addition to the actual informed consent for the intervention, extensive clarification of existing contradictory information is required.

The aim of this research project is to survey pregnant patients prior to receiving an anaesthesiological consultation about their previous knowledge of the intended procedure by conducting an anonymous online survey.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women prior to delivery

Exclusion Criteria:

* Women under 18 years of age

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women prior to delivery
Study Population: Pregnant women before delivery for whom a neuroaxiual procedure for pain reduction during childbirth would theoretically be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Preliminary information on neuroaxial analgesic procedures for childbirth | Between the 25+0 week of pregnancy and delivery
  Is prior information available.[yes/no]
Is the prior information based on internet sources? | Between the 25+0 week of pregnancy and delivery
  Is prior information available based on a internet sources.[yes/no]

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
This is not possible without major restrictions due to state, national and european data protection legislation.